CLINICAL TRIAL: NCT02425189
Title: National Long QT Syndrome Registry: Canadian Genetic Heart Rhythm Network |Research Data Registry and Bio Bank
Brief Title: The Canadian National Long QT Syndrome Registry
Acronym: LQTSREG
Status: Completed | Type: Observational
Sponsor: Andrew Krahn (Other)
Responsible Party: Sponsor-Investigator, Andrew Krahn, Professor of Medicine and Head UBC Division of Cardiology, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H14-02344
Record Dates: First submitted 2014-11-13; First posted 2015-04-23 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood Samples drawn:
  1 X 9 ml EDTA
  Samples for bio banking will be stored long-term
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LQT Positive (Group 1): * Gene-positive LQTS patients
  * Gene negative LQTS patients with confirmed phenotypic diagnosis of LQTS (Schwartz score ≥4)
- Asyptomatic Patients (Group 2): Asymptomatic patients, those free of syncope on beta blocker, or gene negative unaffected family members

SUMMARY:
The NLQTS Research Network team aims to build a Canadian collaboration of dedicated investigators that will create a new paradigm in the modern investigation of patients with LQTS and in the description of a new disease modifier.

The project aims to describe the natural history of familial Long QT Syndrome to identify:

1. Low risk patients that do not require protective beta-blocker therapy
2. High-risk patients that require protective beta-blocker therapy and may benefit from a primary prevention ICD. This cohort would contain treated pre-symptomatic individuals effectively protected from harm.

DETAILED DESCRIPTION:
Methods Patients with positive LQTS diagnosis and their family members reviewed in collaborating Canadian Inherited Arrhythmia Clinics will be invited to participate in the registry.

Optional bio bank donation will be offered. Consenting participants will have blood work drawn in their local outpatient laboratory.

Bio banking at other collaborating centres will be done only at centres that have their own bio banking facility at the site investigator's discretion. There will be no central bio banking on a national basis at this time for this project.

Optional Post Mortem Consent:

The next of kin (NOK) may provide consent to include the healthcare information of the deceased family member into the data registry. The NOK may also consent to the storage of any post mortem tissue not required for clinical testing to be stored in the bio bank for future research.

Data Collected Clinical data will be collected from willing/consented registry participants. Their healthcare information will be coded in compliance with Tri Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code that does not use personal information such as the participant's birth day (month and year will be included), health number, social insurance number or name/initials. The coded data will be transferred into the research database.

The master list of registry participants with their study identifiers will be kept separately from the research database. This master list will be stored in an encrypted file within the research office of each site investigators under their supervision. Only the site investigators and their local research staff will have access to this list. The inherited nature of these conditions makes the master list an important and very sensitive document. It will be very important that this list is maintained so that participants may be contacted and informed of any new findings the research may reveal that may affect themselves and their family members.

All medical information pertaining to the cardiac history of inherited arrhythmia patients will be collected. This may include:

* Clinical information
* All diagnostic test results
* Genetic screening results
* Pedigree
* Medications
* Treatments
* Ethnicity

Participants will continue to have their data collected for the research database throughout the entirety of the study. Participants will be able to decline further participation in the registry at any time. The Research Steering Committee will review the data registry annually to assess the integrity of the data and the usefulness of continued data collection. They will also review related research projects that the data may be useful for.

The registry will not contain stored images graphics, test results or reports that would permit identification of individual subjects. The registry may contain procedural images but these will be coded per TCPS criteria as previously described for the participants' data and biological samples.

Follow-up: Patients will be followed based on severity of presentation (previous cardiac arrest or arrhythmic syncope, or family cascade screening). Vital status(cadiac events) will be determined in person or by telephone annually in all patients enrolled. As per standard care, participants with previous cardiac arrest or arrhythmic syncope on beta-blockers will be followed in person every 12 months (Group 1), and asymptomatic patients, those free of syncope on beta blocker, or gene negative unaffected family members (Group 2) every 2 years (or at the discretion of the site investigator). An annual resting ECG is possible for all participants, and exercise testing will be repeated every 2 years in Group 1, and every 3-4 years in Group 2 based on the clinical practice of the enrolling centre.

Research Database The database will be hosted on the University of British Columbia Research Server. This research institute is in compliance with National Canadian/Provincial PIPEDA privacy guidelines. Data will be entered directly into the e-CRFs for electronic submission to a password protected internet-based server located at the University of British Columbia Research DNS: cio.ciahealth.org IP Address: 142.103.184.100 Server: UBCIT Virtual Server Location: UBC University Data Center (UDC) Pharmaceutical Sciences Building 2405 Wesbrook Mall, Vancouver, BC V6T1Z3 Institute, housed on the Kelowna BC campus and will not collect any personal identifiers.

Individual subject medical information obtained as a result of this registry is considered confidential and disclosure to third parties is prohibited except for the following reason: relevant medical information may be given to the subject's personal physician or to other appropriate medical personnel responsible for the participant's welfare.

Bio Bank Biological samples will be coded in compliance with Tri Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code that does not use personal information such as the participant's birth date, health number, social insurance number or name/initials. The coded biological samples will be stored in the James Hogg Research Centre at St. Paul's Hospital in Vancouver, British Columbia. The coded samples will be linked to the master list kept securely in the research office of the collaborating site investigators. Only site investigators and their local research staff will have access to the master list.

Blood Samples drawn:

1 X 9 ml EDTA

Samples for bio banking will be stored long-term in the James Hogg Research Centre (JHRC) Bio Bank at St. Paul's Hospital in Vancouver for future research. Specimens will be stored in -20 and -80 degree freezers located in a secure area within the JHRC. The freezers are in a dedicated, electronically monitored room managed by JHRC. Inventory management will include retrieving samples, reporting inventory and sample history, and tracking samples with FreezerWorks Unlimited software.

Post mortem samples not required for clinical purposes may be stored in the Bio Bank for future research. In these cases, the sample will be used for research only if the NOK is in agreement to the use of the sample. The investigators will be responsible for notifying the NOK if the sample is to be relocated and for what purpose this is proposed. Written documentation of the notification and consent to proceed from NOK will be required. The NOK will be responsible for keeping the enrolling centre up to date with their contact information so that contact for future use of the sample is feasible. The investigators will be diligent in their attempt to notify the NOK but this may not be feasible in all cases.

Database/bio bank access and Oversight Dr. Andrew Krahn will have ultimate responsibility for the database/bio bank. Investigators wishing to access and use certain data/specimens from the registry/bio bank will submit requests to Dr. Krahn and the Steering Committee for review and approval. Institutional ethics review and approval will be required for new projects. Projects other than retrospective data review will need to seek informed consent from the participant before the data can be extracted from the database.

The National Long QT Syndrome Registry and Bio bank Research Steering Committee The Steering Committee (SC) will be responsible for the design, execution, analysis, and reporting of the study, and will assign appropriate responsibilities to the other study committees. The SC will monitor study progress, execution and management. The SC will be comprised of the Principal Investigator (Chair), who will be the Data/Bio Specimen Steward, and all co applicants. The team is composed of adult electrophysiologists (EPs) that oversee inherited arrhythmia clinics (Drs. Martin Gardner, Hank Duff, Jeff Healey, Jason Roberts, Andrew Krahn, Zach Laksman, Collette Seifer, Mario Talajic, Rafik Tadros, Paul Angaran, Christian Steinberg, Martin Green, Richard Leather, Shane Kimber), and 4 counterpart pediatric EPs (Robert Hamilton, Shubhayan Sanatani, Joseph Atallah, Anne Fournier). The SC will generate an annual report outlining the study's contributions to the scientific community and usefulness of the data . A formal Data and Safety Monitoring Committee will not be created because this is a registry without planned therapeutic comparative studies.

Requests for future use and sharing of the data/specimens will be evaluated according to the following criteria:

* The objectives and hypothesis of the proposed research in relation to established and emerging basic and clinical science
* The proposed research's scientific, clinical and medical importance and translational potential
* Commitment to provide a publication or presentation copy of the primary research data to supplement or complement the registry information
* The proposed test's or research's unique nature and the importance of its validation in LQTS
* The proposed research's duration, demographics, patient population, health economic situation, and probability of success
* Whether the potential benefits and application are local or international in scope
* The quantity of study data required and the commitment to reimburse the full cost associated with delivery of study data
* The contribution that the applicant has made to the registry

Data/Specimen Sharing In addition to the research carried out by the Study Team, some data/specimens may be shared with researchers at other universities; only aggregate coded data would be released for these purposes. These data/specimens may be used by a variety of sources. Prior to data/specimen release, the SC will review written request for access. It is anticipated that there may be requests to pool de-identified data/specimens with data/specimens from other Canadian or international registries/banks in order to answer investigator initiated questions about patient selection, rare events, and long term outcomes.

Statistical Analysis At this phase there is no planned statistical analysis. Descriptive analysis will be performed on the entire cohort, and standard statistical approaches will be used. The current REB application is focused on the permission to prospectively collect data/specimens from the participants and to store it in a coded repository.

Ethical Considerations Participants in this project will be aware that they may not hear any individual results about their own (or deceased NOK's) research data or bio specimen. However, it is possible that there may be future research findings that the investigators may be obliged to inform the individual participants about. These would include findings affecting the heart health of the participant and/or their first-degree family members. Participants will be aware that they may be contacted in the future if there are findings that may affect their heart health care.

Future Research This national approach to case finding and management represents a step towards a population-based approach to studying a "rare" disease (1:2500). The knowledge translation strategy aims to enhance public and health care professional awareness of warning signs, deliver structured histories to assess risk, and improve ECG interpretation skills. This will be imperative to begin a health system approach to recognition of LQTS.

ELIGIBILITY:
Inclusion Criteria:

1. All age groups will be included
2. Gene-positive LQTS patients
3. Gene negative LQTS patients with confirmed phenotypic diagnosis of LQTS (Schwartz score ≥4)
4. Genotype- or phenotype- negative family members of gene- or phenotype- positive LQTS patients evaluated as part of family screening (cascade screening)
5. Informed and willing consent

Exclusion:

1. Geneotype- and phenotype-negative patients without an affected family member 2 .Unwilling or unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with positive LQTS diagnosis and their family members reviewed in collaborating Canadian Inherited Arrhythmia Clinics will be invited to participate in the registry.
  Optional bio bank donation will be offered. Consenting participants will have blood work drawn in their local outpatient laboratory.
Sampling Method: Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2014-11; Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Natural Course of Long QT | Three Years
  Changes to diagnosis, medications, treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krahn, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada